CLINICAL TRIAL: NCT05722041
Title: Soft Tissue Volume Changes in the Posterior Area With Socket Sealing Abutment. Randomized Controlled Trial.
Brief Title: Soft Tissue Volume Changes in Posterior Socket Sealing Abutment.
Status: Active, not recruiting | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: CUSTOM
Record Dates: First submitted 2022-08-11; First posted 2023-02-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dental Implants
Keywords: Dental implant; Immediate implants; Custom Abutment; Sealing Socket Abutment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Customized Abutment: Customized abutment will be placed after molar immediate implant placement.
  Interventions: Procedure: Immediate dental implant placement
- Conventional Abutment: Conventional abutment will be placed after molar immediate implant placement.
  Interventions: Procedure: Immediate dental implant placement

INTERVENTIONS:
Procedure: Immediate dental implant placement — Placement of one dental implant immediately after tooth extraction.
  Other Names: Dental implant surgery

SUMMARY:
The aim is to clinically evaluate the effect of the alveolar sealing technique using a customised abutment on soft tissue volume changes following molar extraction and immediate dental implant placement.

DETAILED DESCRIPTION:
A sample of 20 patients in ASAI health status who agree to be involved in the study after giving their consent and who require immediate post-extraction implant treatment in the molar area will be recruited.

The soft tissue status before and 6 months after tooth extraction will be recorded by means of a digital impression taken with the same intraoral scanner.

The patient will be asked to complete a 7-question questionnaire to inform us about his or her perception of the therapeutic process and the final result.

A comparative volume measurement will be made by digitally superimposing the two mesh files obtained before and 6 months after the treatment.

Statistical data will be analysed by an external statistician and conclusions will be drawn about the effect of the technique on soft tissue volume as well as the patient's perception of the procedure and its outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients ASA I
* Need for molar postextraction immediate implant

Exclusion Criteria:

* When the cortical bone is affected and the alveolus presents bone deficiencies
* When dental implant may not be placed due to medical conditions

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are assisted in private dental office.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue dimensional changes | From 0 to 6 months
  The changes that occur in the soft tissues in millimetres by comparing the digital impressions before and 6 months after the treatment using specific software.

SECONDARY OUTCOMES:
Patients satisfaction | From 0 to 6 months
  Patients will be asked about their satisfaction after the treatment in a Numerical Rate Scale form 0 (Not satisfied) to 10 (Very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, PhD, Principal Investigator — Clinica Dental Esteve
Locations (1):
- Clínica Dental esteve, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data sets obtained during the course of this study will be made available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Chu SJ, Salama MA, Garber DA, Salama H, Sarnachiaro GO, Sarnachiaro E, Gotta SL, Reynolds MA, Saito H, Tarnow DP. Flapless Postextraction Socket Implant Placement, Part 2: The Effects of Bone Grafting and Provisional Restoration on Peri-implant Soft Tissue Height and Thickness- A Retrospective Study. Int J Periodontics Restorative Dent. 2015 Nov-Dec;35(6):803-9. doi: 10.11607/prd.2178. PMID 26509983
- [Background] Finelle G, Lee SJ. Guided Immediate Implant Placement with Wound Closure by Computer-Aided Design/Computer-Assisted Manufacture Sealing Socket Abutment: Case Report. Int J Oral Maxillofac Implants. 2017 Mar/Apr;32(2):e63-e67. doi: 10.11607/jomi.4770. PMID 28291855
- [Background] Ruales-Carrera E, Pauletto P, Apaza-Bedoya K, Volpato CAM, Ozcan M, Benfatti CAM. Peri-implant tissue management after immediate implant placement using a customized healing abutment. J Esthet Restor Dent. 2019 Nov;31(6):533-541. doi: 10.1111/jerd.12512. Epub 2019 Jul 3. PMID 31268244
- [Background] Conejo J, Atria PJ, Hirata R, Blatz MB. Copy milling to duplicate the emergence profile for implant-supported restorations. J Prosthet Dent. 2020 May;123(5):671-674. doi: 10.1016/j.prosdent.2019.05.035. Epub 2019 Oct 1. PMID 31582167
- [Background] Alexopoulou M, Lambert F, Knafo B, Popelut A, Vandenberghe B, Finelle G. Immediate implant in the posterior region combined with alveolar ridge preservation and sealing socket abutment: A retrospective 3D radiographic analysis. Clin Implant Dent Relat Res. 2021 Feb;23(1):61-72. doi: 10.1111/cid.12974. Epub 2021 Jan 13. PMID 33438320
- [Background] Lilet R, Desiron M, Finelle G, Lecloux G, Seidel L, Lambert F. Immediate implant placement combining socket seal abutment and peri-implant socket filling: A prospective case series. Clin Oral Implants Res. 2022 Jan;33(1):33-44. doi: 10.1111/clr.13852. Epub 2021 Oct 22. PMID 34551159
- [Background] Perez A, Caiazzo A, Valente NA, Toti P, Alfonsi F, Barone A. Standard vs customized healing abutments with simultaneous bone grafting for tissue changes around immediate implants. 1-year outcomes from a randomized clinical trial. Clin Implant Dent Relat Res. 2020 Feb;22(1):42-53. doi: 10.1111/cid.12871. Epub 2019 Dec 3. PMID 31797548
- [Background] Fernandes D, Nunes S, Lopez-Castro G, Marques T, Montero J, Borges T. Effect of customized healing abutments on the peri-implant linear and volumetric tissue changes at maxillary immediate implant sites: A 1-year prospective randomized clinical trial. Clin Implant Dent Relat Res. 2021 Oct;23(5):745-757. doi: 10.1111/cid.13044. Epub 2021 Aug 22. PMID 34423560